CLINICAL TRIAL: NCT07106073
Title: La Febbre Nelle Cure Palliative
Brief Title: Fever In Palliative Care
Status: Completed | Type: Observational
Sponsor: Stefania Cheli (Other)
Responsible Party: Sponsor-Investigator, Stefania Cheli, Study coordinator, ASST Fatebenefratelli Sacco
Organization: ASST Fatebenefratelli Sacco (Other)
Other Study IDs: La febbre
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Fever; Palliative Care; Terminal Illness
Keywords: Fever; Palliative Care; Hospice Care; Terminally ill patients; Infectious Diseases Hospice
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of demographic, anthropometric and clinical data. — Data collected is:
  * demographic data: age, sex;
  * anthropometric data: weight, height, body mass index;
  * clinical data:
    * Palliative Performance Scale;
    * Palliative Prognostic Index;
    * comorbidities;
    * therapy;
    * presence of medical devices;
    * presence of pressure injuries;
    * time on waiting list;
    * place of care;
    * primary diagnosis;
    * length of stay;
    * symptom burden at admission (Edmonton Symptom Assessment System);
    * onset of fever and its characteristics (duration, intensity, treatment, etiology);
    * need for sedation (duration, refractory symptom(s));
    * outcome.

SUMMARY:
The goal of this observational study is to evaluate the frequency and characteristics of fever in terminally ill adult patients admitted to the Infectious Diseases Hospice at Luigi Sacco Hospital in Milan. The main questions it aims to answer are:

* How often does fever occur in terminally ill patients during hospice care?
* What are the typical features of fever in this population in terms of intensity, duration, possible causes, and treatment strategies?
* Is there any correlation between the occurrence of fever and patients' clinical characteristics, such as age, sex, BMI, comorbidities, and palliative prognostic scores (PPS and PPI)?

Participants will be adult patients (≥18 years) with a life expectancy of more than 24 hours and less than 3 months.

During their stay, the following data will be collected:

* Presence and characteristics of fever (temperature, duration, treatment, suspected cause)
* Clinical and demographic information (e.g., age, sex, BMI, comorbidities, performance status)
* Details on hospitalization (e.g., symptom burden, need for palliative sedation, outcome)

The study will enroll approximately 250 patients consecutively over a 48-week period. No additional procedures or treatments beyond standard clinical care will be required.

DETAILED DESCRIPTION:
Fever is a common clinical finding in palliative care, but its prevalence, causes, and management in terminally ill patients remain poorly documented. Existing studies report highly variable frequencies of fever near the end of life, ranging from 3% to 24%, depending on the population and setting. In this context, understanding the patterns and implications of fever in hospice patients is critical to improve symptom management and guide clinical decision-making.

This prospective, non-profit, single-center cohort study aims to collect real-world data on the presence of fever in a terminal population admitted to the Infectious Diseases Hospice at Luigi Sacco Hospital in Milan. The study will prospectively collect clinical, demographic, and treatment-related variables over a continuous 48-week period, without any deviation from routine clinical practice. By examining associations with prognostic indices, comorbidities, and symptom burden, the study also seeks to clarify whether fever represents a relevant marker of disease trajectory or end-of-life decline.

Data will be analyzed in aggregated, de-identified form using both descriptive and inferential statistics. This study is expected to contribute to filling a knowledge gap in palliative care literature and may help develop evidence-based guidance for the diagnostic and therapeutic management of fever in hospice settings.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients;
* Age ≥ 18 years;
* Terminally ill patients with an estimated life expectancy between 24 hours and 3 months;
* Signed informed consent.

Exclusion Criteria:

* Patients under 18 years of age;
* Terminally ill patients with a life expectancy < 24 hours
* Non-terminal patients admitted for respite care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Hospice of Infectious Diseases at Luigi Sacco Hospital, ASST Fatebenefratelli Sacco, Milan, Italy. The study population includes adult terminally ill patients admitted for end-of-life care.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Frequency of Fever in Terminally Ill Patients | 48 weeks
  Number of patients who develop at least one febrile episode (defined as body temperature >37.5°C) during their stay in the hospice.
  Unit of Measure: Number of patients

SECONDARY OUTCOMES:
Intensity of Fever | 48 weeks
  Maximum temperature recorded during febrile episodes among patients who develop fever.
  Unit of Measure: Degrees Celsius (°C)

OTHER OUTCOMES:
Duration of Fever | 48 weeks
  Number of consecutive days with fever for each febrile episode. Unit of Measure: Days
Clinical Correlates of Fever | 48 weeks
  Association between fever occurrence and clinical/demographic factors including age, sex, BMI, comorbidities, Palliative Performance Scale (PPS), and Palliative Prognostic Index (PPI).
  Unit of Measure: Odds Ratios or correlation coefficients (as per analysis plan)
Length of Stay in Hospice | 48 weeks
  Number of days each patient remained in hospice care before discharge or death. Unit of Measure: Days
Etiology and Management of Fever | 48 weeks
  Presumed clinical cause of fever (e.g., infection, neoplastic fever) and therapeutic approach (e.g., antibiotics, antipyretics, supportive care).
  Unit of Measure: Number of patients per etiology and management category
Symptom Burden at Admission | At admission
  Assessment of physical and psychological symptom severity at admission using the Edmonton Symptom Assessment System (ESAS). Each symptom is rated on a scale from 0 (none) to 10 (worst possible).
  Unit of Measure: ESAS scores per symptom (0-10)
Palliative sedation | 48 weeks
  Number of patients who required palliative sedation during their hospice stay. Unit of Measure: Number of patients
Patient Outcome at End of Stay | 48 weeks
  Status at the end of hospice stay (discharged or deceased in hospice). Unit of Measure: Number of patients per outcome category
Place of Care Before Admission | At admission
  Care setting prior to hospice admission (e.g., home, hospital, nursing facility).
  Unit of Measure: Number of patients per care setting category
Clinical and Demographic Characteristics at Admission | At admission
  Baseline characteristics including:
  * Age (years)
  * Sex (male/female)
  * Primary diagnosis (e.g., cancer, HIV, neurodegenerative diseases)
  * Comorbidities (as per clinical records)
  * Functional status using the Palliative Performance Scale (PPS)
  * Prognosis using the Palliative Prognostic Index (PPI) Unit of Measure: Descriptive statistics (e.g., mean, median, frequency)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No